CLINICAL TRIAL: NCT01943773
Title: Functional Prehabilitation and Major Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1590
Record Dates: First submitted 2013-08-12; First posted 2013-09-17 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Surgical Complication; Physical Therapy; Timed Up and Go
Keywords: delirium; surgery; operation; geriatric; complication
MeSH Terms: conditions — Delirium | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): The intervention will consist of nine 45 minute long physical therapy sessions. Sessions will occur three times weekly at the patient's home.
  Interventions: Procedure: Functional Assessment; Procedure: Prehabilitation
- No Prehabilitation (Experimental): The control group will undergo routine pre-operative management.
  Interventions: Procedure: Functional Assessment

INTERVENTIONS:
Procedure: Functional Assessment — Both arms of the study will undergo functional assessments at three points during the study progress.
  BASELINE ASSESSMENT: On study entry, each participant will have a timed up-and-go, Mini Mental Status Exam, de Morton, Modified Physical Performance Test (MPPT), and a short physical performance battery performed.
  ASSESSMENT OF INTERVENTION EFFECTIVENESS:
  Immediately prior to the operation, all participants will undergo repeat testing. The difference in scores between the preoperative assessment and the initial assessment at enrollment will be compared in the control and intervention groups.
  POST-OPERATIVE ASSESSMENT: Repeat testing will be performed 60 days following the operation.
Procedure: Prehabilitation — The intervention will consist of nine 45 minute long physical therapy sessions.
  Arms: Prehabilitation

SUMMARY:
Purpose: To compare post-operative functional outcomes in patients undergoing preoperative functional prehabilitation versus standard of care preoperative management in older adults undergoing major elective operations.

Hypothesis: Older adults undergoing preoperative functional prehabilitation (nine sessions of home physical therapy over three weeks) will have improved physical function and reduced delirium in comparison to usual preoperative care following major abdominal and thoracic operations.

Specific Aims:

(#1) To compare the difference in the timed up-and-go, Mini Mental Status Exam (MMSE), the de Morton Mobility Index, Modified Physical Performance Test (MPPT), and short physical performance battery scores in the control and intervention groups at the preoperative and initial assessment timepoints.

(#2) To compare the difference in the timed up-and-go, Mini Mental Status Exam (MMSE), the de Morton Mobility Index, Modified Physical Performance Test (MPPT), and short physical performance battery scores in the control and intervention groups at the 60-days postoperative and the initial assessment timepoints.

(#3)To compare the rates of ICU delirium and need for post-discharge institutionalization in patients in the control and interventions groups.

(#4) To compare post-operative complications

DETAILED DESCRIPTION:
BACKGROUND Prehabilitation has been studied in relation outcomes after surgery. One common area studied is how it affects post-operative outcome for knee replacement patients. Prehabilitation was found to increase strength and function in older adults. {Swank, 2011. #1} Prehabilitation increased leg strength and the ability to perform functional tasks in these patients.

Prehabilitation has also been studied in patients undergoing coronary artery bypass graft surgery (CABG). Primary outcome measures were: anxiety and length of hospital stay; secondary outcome measures were: depression, physical functioning, cardiac misconceptions and cost utility. Prehabilitation was found to decrease depression and improve physical functioning. {Furze, 2009. #2}

Prehabilitation was also found in one study to reduce postoperative complications, length of stay, and declines in functional disability compared to the control group, while improving quality of life, in patients having cardiac and abdominal surgery. {Carli, 2005. #3}

No research has been done linking prehabilitation to the incidence of delirium. The research team has extensive experience studying delirium. Decreased cognition and functional ability has been linked to delirium and poorer outcomes post-operatively. {Robinson, 2009. #4}. Theoretically, by improving functional ability pre-operatively, post-operative outcomes will improve and delirium will decrease. This study will examine if this is true.

The current standard of care for abdominal and non-cardiac thoracic operations does not involve prehabilitation. (Cardiac operations were excluded due to the increased risk for heart-related complications during prehabilitation, such as Myocardial Infarction (MI).) The control group will receive standard of care pre-operative care, with the exception of baseline functional assessments.

OUTCOME MEASURES:

Primary Outcome Variable: A timed up-and-go, Mini Mental Status Exam, the de Morton Mobility Index, Modified Physical Performance Test (MPPT), and a short physical performance battery will be performed 60 days following the operation. The difference in the timed up-and-go and the short physical performance battery between 60 days postoperatively and at the initial assessment will be compared in the control and intervention groups.

Secondary Outcomes: The secondary outcome variables will be the rate of need for discharge to an institutional care facility and ICU delirium. These two variables will be compared in the control and intervention groups.

Other Outcomes: Evaluate post-operative complications. These two variables will be compared in the control and intervention groups.

STUDY DESIGN AND RESEARCH METHODS Baseline Assessment: On study entry, each participant will have a timed up-and-go, Mini Mental Status Exam, de Morton, Modified Physical Performance Test (MPPT), and a short physical performance battery performed. Routine demographics will be performed. Traditional and geriatric preoperative variables will be recorded.

Study Groups: Participants will be randomized to receive standard of care (control) or the intervention of prehabilitation.

1. Control Group: The control group will undergo routine pre-operative management.
2. Intervention Group: The intervention will consist of nine 45 minute long physical therapy sessions. Sessions will occur three times weekly at the patient's home.

Assessment of Intervention Effectiveness: Immediately prior to the operation, all participants will undergo repeat timed up-and-go, Mini Mental Status Exam, the de Morton Mobility Index, Modified Physical Performance Test (MPPT), and short physical performance battery. The difference in scores between the preoperative assessment and the initial assessment at enrollment will be compared in the control and intervention groups.

Operations: The scheduled operation will be performed.

Postoperative Adverse Outcomes: Postoperative adverse outcomes will be recorded using standardized definitions.

DATA ANALYSIS PLAN A sample size of 100 people, because we anticipate many will complete the Up and Go in 10 seconds and faster and will be screen fails. A total of 40 subjects will be randomized, 20 per group. The outcomes of timed up and go, Short Physical Battery, Modified Physical Performance Test (MPPT), and de Morton will be compared from baseline to immediately pre-operatively and immediately post-operatively.

The data will be compared as continuous variables using a non-parametric T-test. Baseline demographic clinical data will be compared in the study and control groups using non-parametric chi square or T-test where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years and older undergoing major abdominal and non-cardiac thoracic operations with an anticipated postoperative ICU stay will be eligible for initial screening. A timed up-and-go assessment will be performed on all who individuals interested in participating. Individuals with a timed up-and-go score of greater than 10 seconds are eligible to participate.
* Women and men will both be recruited for the study. Minorities and non-minorities will be recruited for the study.

Exclusion Criteria:

* Participants under 50 years
* Patients not going to the ICU post-operatively
* Patients having a different kind of operation than major abdominal/non-cardiac thoracic
* Those who complete the timed up-and-go in 10 seconds or less or
* patients who cannot complete the timed up-and-go
* Patients who cannot undergo informed consent
* Patients with vision impairments who cannot visualize the pictures involved with the CAM-ICU
* Patients who do not speak English will be excluded so that confusion created by a language barrier is not confused with post-operative delirium.
* Pregnant women, prisoners, and decisionally challenged subjects.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Post-operative Functional Assessment | 60 days post-operatively
  Timed up-and-go score 60 days post operatively.

SECONDARY OUTCOMES:
Discharge status | Discharge from hospital, expected to be 7 days
  The secondary outcome variable will be the rate of need for discharge to an institutional care facility. This variables will be compared in the control and intervention groups.
Post-operative complications | 30 days post-operatively
  The incidence of post-operative complications, including delirium, will be examined.
Functional and mental battery scores postoperatively | 60 days postoperatively
  A timed up-and-go, Mini Mental Status Exam, the de Morton Mobility Index, Modified Physical Performance Test (MPPT), and a short physical performance battery will be performed 60 days following the operation. The difference in the timed up-and-go and the short physical performance battery between 60 days postoperatively and at the initial assessment will be compared in the control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Robinson, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Denver Veterans Affairs Medical Center, Denver, Colorado

REFERENCES:
- [Background] Swank AM, Kachelman JB, Bibeau W, Quesada PM, Nyland J, Malkani A, Topp RV. Prehabilitation before total knee arthroplasty increases strength and function in older adults with severe osteoarthritis. J Strength Cond Res. 2011 Feb;25(2):318-25. doi: 10.1519/JSC.0b013e318202e431. PMID 21217530
- [Background] Furze G, Dumville JC, Miles JN, Irvine K, Thompson DR, Lewin RJ. "Prehabilitation" prior to CABG surgery improves physical functioning and depression. Int J Cardiol. 2009 Feb 6;132(1):51-8. doi: 10.1016/j.ijcard.2008.06.001. Epub 2008 Aug 15. PMID 18703241
- [Background] Carli F, Zavorsky GS. Optimizing functional exercise capacity in the elderly surgical population. Curr Opin Clin Nutr Metab Care. 2005 Jan;8(1):23-32. doi: 10.1097/00075197-200501000-00005. PMID 15585997
- [Background] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695